CLINICAL TRIAL: NCT03241667
Title: Blood Flow Effects on Silicon Substrates
Status: Withdrawn | Type: Observational
Why Stopped: IRB application withdrawn
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: AK2017
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood testing, hemocartridge system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: HemoCartridge — Our goal is to apply MEMS (microelectromechanical systems) and nanotechnology to miniaturize the bioartificial kidney (BAK) into an implantable, self-monitoring, and self-regulating renal surrogate. The implantable BAK (iBAK) is a biocompatible cartridge containing stacks of hemofilter membranes (HemoCartridge) and renal tubule cell bioreactors (BioCartridge) combined to mimic nephron function. Here, we plan to test ONLY the material being used to construct the HemoCartridge, to be sure in humans when substituted for a standard hemodialysis filter, subjects don't develop any clinical problems or side effects during several hours of blood exposure to the material. The AK material will be engineered by the study team to allow the system to be substituted in place of a standard HD filter.

SUMMARY:
This is a non-randomized, open label, uncontrolled first in human safety study, testing the the material used in the artificial kidney device in subjects already on hemodialysis.

Six subjects already on hemodialysis, who meet the study inclusion and exclusion criteria, and who dialyze at one of the UCSF associated hemodialysis units will be recruited. Each subject will be tested during one non hemodialysis day, at the UCSF Moffitt-Long Hospital Acute Hemodialysis Unit (AHU).

The artificial kidney engineers have created a blood flow system that can be substituted for the dialysis filter in a standard hemodialysis machine. This is NOT a dialysis filter. It allows the subjects blood to come in contact with the material while the blood is being circulated as is regularly done during a hemodialysis session.

DETAILED DESCRIPTION:
For patient safety, the investigators will measure the following labs:

Blood tests (routine safety and frequency). CBC/platelets: q 1 hr, at HD next day ABGs, including lactate: Q 1 hr x 6 Na, K, Cl, Bicarb, BUN, Creatinine, Ca, ionized Ca, Mg, Phos: Start, end, at HD next day Liver function test: Start, end, at HD next day LDH: Start, end, at HD next day Direct Coombs' Test: Start, end, at HD next day ESR and hsCRP: Start, end, at HD next day CPK: Start, end PT/PTT: Start, end

The investigators will also be doing research blood testing:

IL-6: Start, end, at HD next day Complement: Start, end, at HD next day Haptoglobin: Start, end, at HD next day Free Hg: Start, end, at HD next day Fibrinogen, D-dimer: Start, end, at HD next day

In addition, the investigators will do material testing after each participant's test is complete.

Material studies after in vivo testing :

Cell and Protein Adhesion Studies:

1. Scanning Electron Microscopy. The SNM will be placed in a solution containing 2% glutaraldehyde (Electron Microscopy Sciences, Fort Washington, PA), 3% sucrose (Sigma Aldrich) and 0.1 M of phosphate buffered saline (PBS) at 4°C and pH 7.4. After 1 hour, the substrates are rinsed twice with PBS for 30 minutes at 4°C and washed with distilled water for 5 minutes. Dehydration is achieved by placing the substrates in 50% ethanol for 15 minutes while increasing the concentration of ethanol to 60%, 70%, 80%, 90%, and finally 100%. Dehydrated samples are then mounted on aluminum stubs, sputter-coated with gold-palladium, and examined using Scanning Electron Microscopy (SEM; Ultra55 FEGSEM, ZEISS, Peabody, MA).
2. Immunohistochemistry. Platelet adhesion and activation are assessed using immunofluorescence staining for the platelet marker, CD41 (Abcam, Cambridge, MA), and blood-clot marker, tissue plasminogen activator (t-PA, Abcam, Cambridge, MA). Platelets are fixed in 4% paraformaldehyde (Fisher Scientific, Waltham, MA) for 15 minutes followed by incubation in 1% bovine serum albumin for 30 minutes to block nonspecific binding. Platelets are double-labeled as follows: substrates were first incubated with primary antibodies (t-PA), diluted 1:50 in PBS for 60 minutes followed by Alexa Fluor 546 donkey anti-mouse antibody (Invitrogen, Carlsbad, CA) diluted 1:100 in PBS for 60 minutes. Finally, the samples are incubated with anti-human CD41 fluorescein isothiocyanate labeled mouse monoclonal antibody diluted 1:300 in PBS for 60 minutes. Images will be acquired per replicate using a Nikon Eclipse Ti-E motorized inverted microscope (Nikon Instruments Inc., Melville, NY) to obtain a total of 12 images per substrate. The fluorescent intensity of the images is quantified using ImageJ.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 y/o
* ESRD on hemodialysis for at least 3 months
* HD access capable of sustaining at least 300 ml/min blood flow
* Hg > 10.0 g
* Able to take aspirin 81 mg/day for a week prior to the study (for those subjects not already on aspirin)
* Able to read, speak and understand English
* Capable of providing signed informed consent
* HD pt at one of the UCSF outpatient HD units

Exclusion Criteria:

* Subjects with active liver, cardiovascular, neurologic or psychiatric diseases
* Subjects with other active medical problems (e.g., cancer undergoing treatment)
* h/o intradialytic or orthostatic hypotension
* h/o thrombosis or on treatment for thrombosis or use of anticoagulants, excluding antiplatelet agents
* h/o active infection or on antibiotics
* h/o active autoimmune diseases or other inflammatory states
* Ongoing alcohol or illegal drug use
* Pregnant
* H/o hemolysis or allergic reactions to any dialyzers
* Anyone who in the opinion of the study doctors is not qualified to be in the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ESRD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
material stability | 6 months
  This is a first in human safety study, testing the safety of the material used in the artificial kidney device in subjects already on hemodialysis.
  Specific aims include:
  Aim 1: To prove that blood does not degrade the material (see study description for details of processes used) 1.a. by evaluating the effect on surface roughness via scanning electron microscopy of the hemocartridge plates
  1. b. by studying the effect on film thickness via scanning electron microscopy and immunohistochemistry for platelet adhesion.
effects of the hemocartridge materials on inflammatory and coagulation factors in blood | 6 months
  Aim 2: To prove that this material is does not induce inflammatory or coagulation effects nor induce hemolysis. The investigators will do this by drawing blood before, during and after the procedure for inflammatory markers and coagulation factors. The investigators will also evaluate whether any evidence of mechanical dysfunction, such as hemolysis occurs during the treatment. See the detailed study description for the listing and timing of the tests.
  1.c. evaluation of mechanical dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Shuvo Roy, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No